CLINICAL TRIAL: NCT03211650
Title: Efficacy of Intra-articular Injection of Combined Hyaluronic Acid and Platelet-rich Plasma in Knee Degenerative Joint Disease
Brief Title: Efficacy of Hyaluronic Acid and Platelet-rich Plasma Combination in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Regen Lab SA (Industry)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Full Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-HA
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hyaluronic acid + platelet-rich plasma (Experimental): Intra-articular injections of hyaluronic acid combined with platelet-rich plasma
  Interventions: Drug: hyaluronic Acid + platelet-rich plasma
- platelet-rich plasma (Active Comparator): Intra-articular injections of platelet-rich plasma
  Interventions: Drug: platelet-rich plasma
- hyaluronic acid (Active Comparator): Intra-articular injections of hyaluronic acid
  Interventions: Drug: hyaluronic acid

INTERVENTIONS:
Drug: hyaluronic Acid + platelet-rich plasma — Intra-articular injections of hyaluronic acid combined with platelet-rich plasma
  Other Names: Cellular Matrix/A-CP HA Kit
  Arms: hyaluronic acid + platelet-rich plasma
Drug: hyaluronic acid — Intra-articular injections of hyaluronic acid
  Other Names: ArthroVisc40
  Arms: hyaluronic acid
Drug: platelet-rich plasma — Intra-articular injections of platelet-rich plasma
  Other Names: RegenKit-BCT-1
  Arms: platelet-rich plasma

SUMMARY:
The purpose of this study is to evaluate the efficacy of intra-articular injections of combined hyaluronic acid and platelet-rich plasma in knee degenerative joint disease in improving joint function and reducing pain.

ELIGIBILITY:
Inclusion criteria:

* Knee pain for 4 months;
* Knee degenerative sign evaluated with X-ray with a Kellgren-Lawrence grade inferior to 3;
* Patients able to understand the study conditions and willing to participate for its entire duration;
* Patients who signed written informed consent.

Exclusion criteria:

* Severe knee osteoarthritis of grade 4;
* Diabetes mellitus;
* Rheumatoid arthritis;
* Ongoing malignancies;
* Certified allergic reactions towards the administered drugs ;
* Malalignment of mechanical axis of the lower limb (varus > 10 °, valgus > 10 °);
* Coagulopathies;
* Severe cardiovascular diseases;
* Ongoing infections;
* Immunodepression;
* Anticoagulants or anti-platelet agents;
* Haemoglobin < 11 g/dl;
* Platelet count < 150,000/mm^3
* Drug addiction;
* Alcoholism;
* Psychiatric disease;
* Pregnancy or breastfeeding.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
WOMAC score | 6 months after the first intra-articular injection
  Comparison of WOMAC total score among three treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Randelli, Professor, Principal Investigator — Azienda Socio Sanitaria Territoriale Centro Specialistico Ortopedico Traumatologico Gaetano Pini - CTO
Locations (2):
- Italy (2):
  - U.O.C. 1a Divisione, Azienda Socio Sanitaria Territoriale Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan, Milan
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan